CLINICAL TRIAL: NCT01692951
Title: Serum Free Fatty Acid Metabolite Biomarkers of Lung Cancer
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, MD, Outcomes Research Consortium
Other Study IDs: 12-306
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer; Biomarkers; Fatty Acids
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood will be sampled for FFA metabolites
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lung adenocarcinoma patients: Serum samples were collected from patients with lung cancer at the time of their diagnosis, prior to the initiation of treatment. Diagnosis of lung adenocarcinoma was based on pathologic analysis.
  Interventions: Other: serum sample
- Control matched to adenocarcinoma: Control subjects without known cancer and aged from 40 to 75 years should meet at least one of the following criteria: (1) current or ex-smoker with at least a 10 pack-year history, (2) a first-degree relative with a history of lung cancer, or (3) a clinical diagnosis of COPD.
  Interventions: Other: serum sample
- Lung squamous cell carcinoma patients: Serum samples were collected from patients with lung cancer at the time of their diagnosis, prior to the initiation of treatment. Diagnosis of lung squamous cell carcinoma was based on pathologic analysis.
  Interventions: Other: serum sample
- Control matched to squamous cell: Control subjects without known cancer and aged from 40 to 75 years should meet at least one of the following criteria: (1) current or ex-smoker with at least a 10 pack-year history, (2) a first-degree relative with a history of lung cancer, or (3) a clinical diagnosis of COPD.
  Interventions: Other: serum sample

INTERVENTIONS:
Other: serum sample — Serum samples from lung cancer patients were collected at the time of their diagnosis, prior to the initiation of treatment. Serum samples of control subjects were collected from a biobank

SUMMARY:
This study aims to evaluate the performance of serum free fatty acids as biomarkers for the identification of lung cancer.

DETAILED DESCRIPTION:
We will compare the concentration of free fatty acids and their metabolites between patients with lung cancer and control pulmonary patients without known cancer. The diagnostic accuracy will be assessed for potential predictors.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 80
* Lung adenocarcinoma with pathological diagnosis
* Lung squamous cell carcinoma with pathological diagnosis
* Control patients should have at least one of the following criteria: (1) current or ex-smoker with at least a 10 pack-year history, (2) a first-degree relative with a history of lung cancer, or (3) a clinical diagnosis of COPD.

Exclusion Criteria:

- Lung cancer patient without serum sample before the initiation of treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient samples are retrieved from the Cleveland Clinic Biobank.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lung Adenocarcinoma Patients | Control Matched to Adenocarcinoma | Lung Squamous Cell Carcinoma Patients | Control Matched to Squamous Cell
Started | 37 | 111 | 18 | 54
Completed | 37 | 111 | 18 | 54
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lung Adenocarcinoma Patients | Control Matched to Adenocarcinoma | Lung Squamous Cell Carcinoma Patients | Control Matched to Squamous Cell | Total
Number analyzed (Participants) | 37 | 111 | 18 | 54 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 65 (6) | 70 (9) | 68 (6) | 66 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 40 | 7 | 24 | 84
  Male | 24 | 71 | 11 | 30 | 136
Smoking status [Number; unit: participants]
  Never | 1 | 3 | 0 | 3 | 7
  Former | 27 | 76 | 15 | 39 | 157
  Current | 9 | 32 | 3 | 12 | 56
Family history of lung cancer [Count of Participants; unit: Participants] | 6 | 21 | 5 | 16 | 48
COPD [Count of Participants; unit: Participants] | 10 | 32 | 5 | 11 | 58
Amount of Cigarette Smoking as Pack-year [Median (Inter-Quartile Range); unit: pack-year] | 40 [25 to 56] | 40 [26 to 56] | 38 [25 to 50] | 39 [24 to 60] | 40 [25 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Compare Concentration of Fatty Acids and Their Metabolites
Description: Biochemical analysis of serum sample was conducted by an investigator who was strictly blinded to cancer status and patient characteristics.
Time Frame: At the time of diagnosis, prior to the initiation of lung cancer treatment
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Lung Adenocarcinoma Patients | Control Matched to Adenocarcinoma | Lung Squamous Cell Carcinoma Patients | Control Matched to Squamous Cell
Number analyzed (Participants) | 37 | 111 | 18 | 54
mg/mL
  Arachidonic Acid | 5.70 [4.62 to 7.74] | 2.95 [2.26 to 4.63] | 4.24 [3.65 to 5.05] | 3.18 [2.43 to 4.45]
  Linoleic Acid | 0.59 [0.46 to 0.73] | 0.34 [0.22 to 0.52] | 0.44 [0.33 to 0.64] | 0.32 [0.23 to 0.42]
  Hydroperoxyoctadecadienoyl phosphatidylcholine | 22.3 [13.1 to 33.3] | 17.9 [12.3 to 23.6] | 18 [16 to 29] | 18 [14 to 24]
  Hydroxyoctadecadienoylphosphatidylcholine | 2.5 [1.9 to 5.5] | 7.1 [3.2 to 13.1] | 4 [2 to 18] | 9 [4 to 16]
  Azelaoyl platelet activating factor | 0.4 [0.3 to 0.5] | 0.5 [0.3 to 0.8] | 0.5 [0.3 to 0.8] | 0.5 [0.3 to 0.8]
  Azelaoyl phosphatidylcholine | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.2]
  C18-lysophospholipid platelet activating factor | 12.7 [8.6 to 15.7] | 16.5 [13.1 to 19.8] | 13 [11 to 14] | 17 [13 to 20]
  C16-lyso-phosphatidylcholine | 8.3 [6.2 to 17.8] | 9.8 [6.6 to 30.6] | 12 [6 to 52] | 13 [7 to 42]
  C16-lysophospholipid platelet activating factor | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
  5-hydroxyeicosatetraenoic acid | 0.05 [0.04 to 0.07] | 0.03 [0.02 to 0.05] | 0.04 [0.03 to 0.05] | 0.03 [0.02 to 0.04]
  11-hydroxyeicosatetraenoic acid | 0.07 [0.03 to 0.11] | 0.03 [0.02 to 0.05] | 0.04 [0.04 to 0.06] | 0.03 [0.02 to 0.04]
  12-hydroxyeicosatetraenoic acid | 0.94 [0.44 to 1.73] | 0.23 [0.13 to 0.57] | 0.42 [0.18 to 0.95] | 0.22 [0.13 to 0.51]
  15-hydroxyeicosatetraenoic acid | 0.02 [0.01 to 0.02] | 0.01 [0.00 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.01]
  9-hydroxyoctadecadienoic acid | 0.56 [0.30 to 0.97] | 0.58 [0.32 to 0.87] | 0.52 [0.36 to 0.68] | 0.51 [0.34 to 0.76]
  13-hydroxyoctadecadienoic acid | 0.43 [0.27 to 0.62] | 0.48 [0.30 to 0.69] | 0.49 [0.38 to 0.73] | 0.44 [0.33 to 0.63]

ADVERSE EVENTS:
Arm/Group | Lung Adenocarcinoma Patients | Control Matched to Adenocarcinoma | Lung Squamous Cell Carcinoma Patients | Control Matched to Squamous Cell
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/111 | 0/18 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/111 | 0/18 | 0/54
Other Adverse Events (participants affected / at risk) | 0/37 | 0/111 | 0/18 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes